CLINICAL TRIAL: NCT01144143
Title: Single Center, Randomized, Double-Blind, Placebo-Controlled Treatment Of Knee Osteoarthritis With Intra-Articular Infliximab
Brief Title: Treatment Of Knee Osteoarthritis With Intra-Articular Infliximab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herbert Lindsley, MD (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Herbert Lindsley, MD, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10702
Record Dates: First submitted 2010-06-10; First posted 2010-06-15 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: Mild to moderate osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Infliximab (Experimental)
  Interventions: Drug: Infliximab
- Salt Water (Placebo Comparator)
  Interventions: Drug: Placebo
- Methylprednisolone acetate (Active Comparator)
  Interventions: Drug: Standard of Care: Methylprednisolone acetate

INTERVENTIONS:
Drug: Infliximab — the study drug will be injected into the joint through a needle
  Arms: Infliximab
Drug: Placebo — the placebo will be injected into the joint through a needle
  Arms: Salt Water
Drug: Standard of Care: Methylprednisolone acetate — Methylprednisolone acetate will be injected into the joint through a needle
  Arms: Methylprednisolone acetate

SUMMARY:
The purpose of this study is to determine if an anti-inflammatory drug, called infliximab, will reduce inflammation in the synovial lining in patients with an early stage of osteoarthritis of the knee. It will also help determine if the study medication decreases the accumulation of synovial fluid and prevents cartilage breakdown.

DETAILED DESCRIPTION:
This is an unbalanced randomized, double-blind pilot study of Infliximab (100 mg), placebo (100 mg) and Methylprednisolone acetate (80 mg). A total of 16 subjects will be randomized; 8 subjects will be randomized to receive infliximab, 4 subjects will be randomized to receive placebo and 4 additional subjects will be randomized to receive Methylprednisolone acetate. Subjects will be seen at screening, day 0, day 14, day 28 and day 56. After study drug injection at day 0, patients will return for follow-up visits at approximately 2 weeks, 1 and 2 months in order to obtain clinical endpoint measures for a total of 10 weeks. Outcome measures include blood tests, MRI, ultrasound, synovial lining tissue biopsy questionnaires and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ age 35 but ≤ age 85.
2. Painful knees for 3-60 months.
3. VAS joint pain score greater than 30 mm (scale 0-100)
4. Knee radiograph showing minimal to moderate change (early OA).
5. No NSAID therapy for at least one week.
6. Have the capacity to understand and sign an informed consent form.
7. Gender: Male or female
8. Women must be postmenopausal (no menstrual period for a minimum of 1 year) or surgically sterilized and have a negative serum pregnancy test on entry in the study. Men must agree to use adequate birth control during the study for 6 months after the infusion of study agent.
9. Men and women of childbearing potential must use adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilization) for the duration of the study and should continue such precautions for 6 months after receiving the last infusion.
10. The screening laboratory test results must meet the following criteria

    1. WBC (white blood cell count): >3.5/uL
    2. Hemoglobin: > 10 gm/dl
    3. Platelets: > 100,000/ul
    4. Serum Creatinine: < 1.8
    5. SGPT (ALT - alanine aminotransferase) <3 times ULN
    6. UA (urinalysis) with microscopic exam: WNL
    7. Negative tests for HbsAg or hepatitis C Ab
    8. PT/PTT: WNL
11. Are considered eligible according to the following TB screening criteria:

    1. Have no history of latent or active TB prior to screening. An exception is made for subjects who have a history of latent TB (defined for the purposes of this study as having had a positive result from either the tuberculin skin test or the QuantiFERON-TB Gold test prior to screening) and documentation of having completed an adequate treatment regimen for latent TB within 3 years prior to the first administration of study agent under this protocol. Adequate treatment for latent TB is defined according to local country guidelines for immunocompromised patients. If no local guidelines for immunocompromised patients exist, US guidelines must be followed. It is the responsibility of the investigator to verify the adequacy of previous anti-TB treatment and provide appropriate documentation.
    2. Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.
    3. Have had no recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to or simultaneously with the first administration of study agent.
    4. Within 1 month prior to the first administration of study agent, either have negative diagnostic TB test results (defined as both a negative tuberculin skin test and a negative QuantiFERON-TB Gold test, as outlined in Attachment 3 and Attachment 4, respectively), or have a newly identified positive diagnostic TB test result (defined as either a positive tuberculin skin test or a positive QuantiFERON-TB Gold test) during screening in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated either prior to or simultaneously with the first administration of study agent. The tuberculin skin test and QuantiFERON-TB Gold test are not required at screening for subjects with a history of latent TB and documentation of having completed adequate treatment as described in Inclusion Criterion 12a. Furthermore, these subjects are not required to initiate additional treatment for latent TB.
    5. Have a chest radiograph (both posterior-anterior and lateral views), taken within 3 months prior to the first administration of study agent and read by a qualified radiologist, with no evidence of current active TB or old inactive TB.

Exclusion Criteria:

1. Moderate to Severe OA, as determined by severe joint space narrowing (Kellgren grade IV) (7) in medial and lateral compartments
2. Insulin-dependent diabetes mellitus.
3. Systemic inflammatory illness, e.g. rheumatoid arthritis.
4. Intra-articular injections within 3 months.
5. Prior treatment with infliximab or other anti-TNF drug.
6. Acute injury to knees (< 2 weeks)
7. Women who are pregnant, nursing, or planning pregnancy within 6 months after the last infusion (this includes father's who plan on fathering a child within 6 months after their last infusion).
8. Have had any previous treatment with monoclonal antibodies or antibody fragments.
9. History of receiving human/murine recombinant products or a known allergy to murine products. A known allergy to murine product is definitely an exclusion criterion
10. Documentation of a positive test for hepatitis B surface antigen or hepatitis C.
11. Have a history of alcohol or substance abuse within the preceding 6 months that, in the opinion of the investigator, may increase the risks associated with study participation or study agent administration, or may interfere with interpretation of results.
12. Have a known history of serious infections (e.g., hepatitis, pneumonia, or pyelonephritis) in the previous 3 months.
13. Have or have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening
14. Currently receiving Coumadin, Ticlid, Plavix, or heparin/heparin analog within 7 days prior to synovial biopsy.
15. Currently receiving aspirin within 7 days prior to synovial biopsy.
16. Have a chest radiograph at screening that shows evidence of malignancy or infection.
17. Have a history of lymphoproliferative disease, including lymphoma or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location (e.g., nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic area), or splenomegaly.
18. Currently have any known malignancy or have a history of malignancy within the previous 5 years, with the exception of basal cell or squamous cell carcinoma of the skin that has been fully excised with no evidence of recurrence as well as carcinoma in situ of the cervix.
19. Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
20. Are unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access.
21. Use of any investigational drug within 30 days prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
22. Presence of a transplanted solid organ (with the exception of a corneal transplant > 3 months prior to screening).
23. Have a concomitant diagnosis or history of congestive heart failure Grade III-IV.
24. Have had a nontuberculous mycobacterial infection or opportunistic infection (e.g., cytomegalovirus, Pneumocystis carinii, and aspergillosis) within 6 months prior to screening.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Lindsley, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University Of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab: Investigational (Infliximab) - 100mg The study drug will be injected into the joint through a needle
- Salt Water: Placebo (Salt Water) - 10 ml Placebo solution will be injected into the joint through a needle
- Methylprednisolone Acetate: Methylprednisolone Acetate (Standard of Care: MPA) - Standard of Care: MPA 80mg injected into the joint through a needle
Period: Overall Study
Arm/Group | Infliximab | Salt Water | Methylprednisolone Acetate
Started | 8 | 4 | 4
Completed | 8 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab | Salt Water | Methylprednisolone Acetate | Total
Number analyzed (Participants) | 8 | 4 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 4 | 15
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 13
  Male | 3 | 0 | 0 | 3
Race/Ethnicity, Customized [Number; unit: Number]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 5 | 3 | 3 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Cellular Infiltrates From Day 0 to Day 28
Description: Cellular infiltration scored 0 to 3
Time Frame: Day 0 to Day 28
Population: In the MPA arm, one subject was excluded from the analysis because their biopsy sample was of insufficient quantity to be processed in the lab.
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab | Salt Water | Methylprednisolone Acetate
Number analyzed (Participants) | 8 | 4 | 3
Participants
  Decreased cellularity | 2 | 0 | 2
  Increased cellularity | 4 | 2 | 0
  Unchanged cellularity | 2 | 2 | 1

2. Secondary Outcome: Change in Joint Effusions From Day 0 to Day 56 Target Knee
Description: Outcome calculated based on Physician observation of joint swelling from 0-3. A score of 0 = no effusion,1 = positive "bulge," 2 = moderate effusion, 3 = tense effusion. The outcome represents the change in means between the two time points.
Time Frame: Change from Day 0 to Day 56
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Salt Water: Placebo (Salt Water) - 10 ml Placebo solution will be injected into the joint through a needlePlacebo: the placebo will be injected into the joint through a needle
Arm/Group | Infliximab | Salt Water | Methylprednisolone Acetate
Number analyzed (Participants) | 8 | 4 | 4
units on a scale | 0.3 (0.5) | 0.0 (0.0) | 0.0 (0.0)

3. Secondary Outcome: Change in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score Target Knee
Description: The WOMAC questionnaire is used to evaluate the condition of patients with osteoarthritis. Patients answer questions based on how they are feeling. The questionnaire has a total of 24 questions which deal with pain, stiffness and physical function. Participants are asked to respond to how difficult it is for them to do/complete an activity. There is a total possible score of 96. A score of 0 equals no difficulty completing any of the 24 activities. A score of 96 would indicate extreme difficulty with all activities.
Time Frame: Change from Day 0 to Day 56
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Normal Saline: Placebo: the placebo will be injected into the joint through a needle
Arm/Group | Infliximab | Normal Saline | Methylprednisolone Acetate
Number analyzed (Participants) | 8 | 4 | 4
units on a scale | -25.9 (18.1) | -9.3 (27.2) | 2.0 (5.8)

4. Secondary Outcome: Change in Levels of Serum IL-6
Time Frame: Change from Day 0 to Day 56
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Infliximab | Salt Water | Methylprednisolone Acetate
Number analyzed (Participants) | 8 | 4 | 4
pg/ml | -0.4 (2.0) | 8.1 (13.0) | 5.5 (9.5)

5. Secondary Outcome: Change in Serum CRP Day 0 to Day 56
Description: Serum measure of systemic inflammation
Time Frame: Day 0 to Day 56
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Infliximab | Salt Water | Methylprednisolone Acetate
Number analyzed (Participants) | 8 | 4 | 4
mg/dl | -0.18 (0.37) | -0.15 (0.30) | 0.08 (0.81)

6. Secondary Outcome: Change in Serum SAA Levels Day 0 to Day 56
Description: Serum Amyloid A
Time Frame: Day 0 to Day 56
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Infliximab | Salt Water | Methylprednisolone Acetate
Number analyzed (Participants) | 8 | 4 | 4
ug/ml | -1.0 (2256) | -715.6 (1043) | -1580.2 (4819)

ADVERSE EVENTS:
Time Frame: Patients were observed for adverse events for 70 days (from screening (Day -14) through Day 56).
Description: Event information collected via subject reporting at visits.
Arm/Group | Infliximab | Salt Water | Methylprednisolone Acetate
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/8 | 1/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=8) | Salt Water (N=4) | Methylprednisolone Acetate (N=4)
Pulled Muscle in Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pulling and Popping Sensation in Knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling in Left Knee Following Biopsy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in Left knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain at Biopsy Site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Twisted Left knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes